CLINICAL TRIAL: NCT03627806
Title: Disparities in Stroke Outcomes and Care Delivery in Patients With Atrial Fibrillation: FLorida Puerto Rico Atrial Fibrillation Stroke Study (FLiPER-AF)
Brief Title: FLorida Puerto Rico Atrial Fibrillation Stroke Study (FLiPER-AF)
Acronym: FLiPER-AF
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Tatjana Rundek, MD, PhD, Principal Investigator, University of Miami
Other Study IDs: CV185-564
Record Dates: First submitted 2018-04-29; First posted 2018-08-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
Keywords: Disparities; Florida-Puerto Rico Stroke Registry
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, FL-PR Stroke Registry will be used to determine novel data on disparities in stroke care and outcomes for patients with Atrial Fibrillation (AF) in 'real life' hospital setting. Investigators will evaluate clinical practice for AF detection and treatment in stroke patients within large stroke hospital systems of care with multi-ethnic patient populations and thereby representative of the states of Florida and Puerto Rico. The results of this study will be of critical importance for secondary stroke prevention by identifying gaps in stroke care for patients with AF and by recognizing the needs for developing targeted interventions to reduce disparities in diverse populations of stroke patients with AF and improve systems of care for all stroke patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* age is 18 and older
* primary diagnosis of ischemic stroke
* enrolled in the Florida - Puerto Rico Stroke Registry

Exclusion Criteria:

* primary diagnosis of intracerebral hemorrhage
* diagnosis of subarachnoid hemorrhage
* stroke not otherwise specified
* no stroke related diagnosis
* admission for elective carotid intervention only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is derived from the Florida-Puerto Rico Stroke Registry to Reduce Stroke Disparities. In-hospital acute stroke performance measures are documented and obtained through the American Heart Association (AHA) Get With The Guidelines-Stroke (GWTG-S) premier hospital quality improvement program and GWTG-S data collection instruments. Through the GWTG-S data, the Registry currently has close to 169,000 patients enrolled since 2010.
Sampling Method: Probability Sample
Enrollment: 104308 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
In-Hospital Quality of Care Acute Stroke Measures | 5 years
  As measured by modified rankin score (mRS) at discharge (a score that measures the degree of disability or dependence in the daily activities of people who have suffered a stroke). A minimum score of 0 indicates no symptoms and therefore no disability. A maximum score of 6 indicates death has resulted

SECONDARY OUTCOMES:
Temporal trends of atrial fibrillation for stroke outcomes | 5 years
  Changes in the occurrence of atrial fibrillation (AF) and its effect on related hospital discharge characteristics among stroke patients
Temporal trends in the frequency of hospital prescriptions at discharge of anticoagulants for stroke patients | 5 years
  Changes over the years measured through the quantification of the frequency hospitals prescribe anticoagulants (i.e., aspirin, warfarin, and novel oral anticoagulants) at discharge
Temporal trends in the frequency of hospital prescriptions for atrial fibrillation monitoring devices | 5 years
  Changes over the years measured through the quantification of the frequency hospitals prescribe atrial fibrillation monitoring devices (i.e., Holter monitoring and prolonged electrocardiogram monitoring).

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Rundek, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sur NB, Wang K, Di Tullio MR, Gutierrez CM, Dong C, Koch S, Gardener H, Garcia-Rivera EJ, Zevallos JC, Burgin WS, Rose DZ, Goldberger JJ, Romano JG, Sacco RL, Rundek T. Disparities and Temporal Trends in the Use of Anticoagulation in Patients With Ischemic Stroke and Atrial Fibrillation. Stroke. 2019 Jun;50(6):1452-1459. doi: 10.1161/STROKEAHA.118.023959. Epub 2019 May 14. PMID 31084325